CLINICAL TRIAL: NCT04779255
Title: Tumescent Anesthesia Interest in Pain Management During a Dynamic Phototherapy (PTD) Session in Vertex Actinic Keratosis Treatment: a Single-center Prospective Randomized Study
Brief Title: Pain Management During a Photodynamic Therapy Session on the Vertex for Actinic Keratosis: Tumescent Anesthesia Interest
Acronym: ANTUKA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-000304-38
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Pain; Actinic Keratosis; Analgesia; Phototerapy; Vertex
MeSH Terms: conditions — Pain; Keratosis, Actinic; Agnosia | interventions — Acetaminophen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tumescent anesthesia (Experimental): Patient who will receive tumescent anesthesia as analgesic treatment
  Interventions: Drug: Procedure (Tumesent anesthesia)
- Painkillers and cold water (Active Comparator): Patient who will receive painkillers 1 hour before photodynamic therapy and cold water during session as analgesic treatment
  Interventions: Drug: Control Arm (Paracetamol)

INTERVENTIONS:
Drug: Procedure (Tumesent anesthesia) — Photodynamic therapy of vertex with a solution of 180 ml of tumescent anesthesia diffused over 1 hour in three different sub-deceasing points.
  Arms: Tumescent anesthesia
Drug: Control Arm (Paracetamol) — Photodynamic therapy of vertex with 1g of paracetamol intake 1 hour before cold water is applied during the session.
  Arms: Painkillers and cold water

SUMMARY:
This study focus on the efficacity of tumescent anesthesia in pain management during a photodynamic therapy on the vertex for treatment of actinic keratosis. To do this we carried out a prospective, randomized, controlled, open-ended study. Our aim is to show a 40% reduction in pain during photodynamic therapy session compared to a conventionally used analgesic method (paracetamol + cold water)

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* Diagnosis of clinical or histological actintic keratoses validated by a dermatologist
* More than 4 vertex actinic keratoses lesions that can be treated with a dynamic phototherapy session
* Free subject, without guardianship or curatorship or subordination
* Person affiliated or beneficiary of a social security plan
* Informed and signed consent by the patient after clear and fair information about the study

Exclusion Criteria:

* Known lidocaine hydrochlostate hypersensitivity, local amide-binding anesthetics or one of the excipients
* Hypersensitivity to paracetamol or one of the excipients
* Weight < 50 kg
* Patients with an elongated TQ interval at the ECG (>450 ms in men and >470 ms in women)
* Patients with recurrent porphyria
* Severe hepato-cellular insufficient patients
* Patients who have received treatment for actinic keratoses in the last three months (cryotherapy, 5-fluorouracil, imiquinod, daylight-PTD)
* Patients who have already participated in this study
* People who do not have a social security plan or do not benefit from it through a third party.
* Persons with enhanced protection, namely minors, persons deprived of their liberty by judicial or administrative decision, persons staying in a health or social institution, adults under legal protection and finally the sick in an emergency situation.
* Pregnant or lactating women, women of childbearing age who do not have effective contraception (hormonal/mechanical: per bone, injectable, transcutaneous, implantable, intrauterine device, or surgical: tubal ligation, hysterectomy, total oophorectomy).
* Concurrent participation in another clinical research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Measure : evaluate the effectiveness of tumescent anesthesia compared to the control group in pain management during a dynamic vertex phototherapy session performed for the management of actinic keratoses. | 8 minutes
  Score of the maximum numerical pain assessment scale from 0 to 10 (0=no pain; 10= pain as bas as can be) felt during the dynamic phototherapy session in both groups.
  This score will be collected at the end of the session.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU, Poitiers, France